CLINICAL TRIAL: NCT00627445
Title: Effect of Biphasic Insulin Aspart 50 Compared to Biphasic Insulin Aspart 30 Both in Combination With Metformin in Chinese Subjects With Type 2 Diabetes
Brief Title: Effect of Biphasic Insulin Aspart 50 on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1858
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 50-50-30 (Experimental): Biphasic insulin aspart 50 administered before breakfast and lunch + biphasic insulin aspart 30 at dinner combined with metformin
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin; Drug: biphasic insulin aspart 50
- BIAsp 30-30 (Active Comparator): Biphasic insulin aspart 30 administered before breakfast and dinner combined with metformin
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Treat-to-target dose titration scheme (dose adjusted individually), s.c. (under the skin) injection before dinner
Drug: metformin — Tablets, 500 - 2000 mg, once, twice or three times daily
Drug: biphasic insulin aspart 50 — Treat-to-target dose titration scheme (dose adjusted individually), s.c. (under the skin) injection before breakfast and lunch
  Arms: BIAsp 50-50-30

SUMMARY:
This trial is conducted in Asia. The trial aims to investigate if the blood glucose control of biphasic insulin aspart 50 is at least as effective as treatment with biphasic insulin aspart 30 both in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with premix human insulin twice daily with or without oral antidiabetic drugs for at least 3 months
* HbA1c (Glycosylated Haemoglobin A1c) between 7.5% - 12.0% (both inclusive)
* FPG (Fasting Plasma Glucose) higher than 7.0 mmol/L
* BMI (Body Mass Index) 23-40 kg/sq.m (both inclusive)

Exclusion Criteria:

* Metformin contraindications according to local practice
* Systemic use of TZDs (thiazolidinediones) for more than 1 month within 6 months prior to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 sites in China
Pre-assignment Details: Eligible subjects were subjects with type 2 diabetes having an HbA1c (Glycosylated Haemoglobin A1c) between 7.5-12.0 %, and treated with premix human insulin twice daily with or without oral anti-diabetic drugs (OADs) for at least 3 months qualifying for an intensified insulin treatment.
Groups:
- BIAsp 50-50-30: Individual adjusted dose of biphasic insulin aspart 50 administered before breakfast and lunch and individual adjusted dose of biphasic insulin aspart 30 at dinner in combination with metformin 500-2000 mg, up to three times daily
- BIAsp 30-30: Individual adjusted dose of biphasic insulin aspart 30 administered before breakfast and dinner in combination with metformin 500-2000 mg, up to three times daily
Period: Overall Study
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Started | 219 | 222
Exposed to Study Drug | 219 | 222
Completed | 210 | 210
Not Completed | 9 | 12
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30 | Total
Number analyzed (Participants) | 219 | 222 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening
  years | 55.5 (8.6) | 55.5 (8.6) | 55.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 113 | 244
  Male | 88 | 109 | 197
BMI [Mean (Standard Deviation); unit: kg/m2] — BMI = Body Mass Index at randomisation
  kg/m2 | 26.06 (2.70) | 26.27 (2.73) | 26.17 (2.71)
Height [Mean (Standard Deviation); unit: cm] — Height at screening
  cm | 162.8 (7.9) | 163.7 (8.4) | 163.2 (8.1)
Weight [Mean (Standard Deviation); unit: kg] | 69.2 (9.8) | 70.5 (9.7) | 69.9 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c)
Description: Change in glycosylated haemoglobin A1c (HbA1c) from week 0 (baseline) to end of treatment (week 16)
Time Frame: week 0, week 16
Population: Intention-to-Treat analysis set (ITT) using LOCF (Last Observation Carried Forward) is all randomised subjects exposed to at least one dose of trial product.
Measure: Least Squares Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 216 | 221
percentage (%) of total haemoglobin | -1.790 (0.057) | -1.517 (0.056)

2. Secondary Outcome: The Percentage of Subjects Achieving HbA1c Treatment Targets
Description: The percentage of subjects who after 16 weeks of treatment met the glycosylated haemoglobin A1c (HbA1c) treatment targets below 7%, or below or equal to 6.5%.
Time Frame: week 16
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 219 | 222
percentage (%) of subjects
  Achieving HbA1c <7.0% | 65 | 52
  Achieving HbA1c <=6.5% | 47 | 29

3. Secondary Outcome: Change and Daily Average in 8-point Plasma Glucose
Description: Change in 8-point plasma glucose from baseline (week 0) to at end of treatment (week 16). 8-point plasma glucose was measured at following time points: Before each meal, 120 minutes after the start of each meal, at bedtime, and at 3:00 AM in the morning. Daily average was calculated at the end of treatment.
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- BIAsp 50-50-30: Individually adjusted dose of biphasic insulin aspart 50 administered before breakfast and lunch in combination with metformin (500-2000 mg up to three times daily)
- BIAsp 30-30: Individually adjusted dose of biphasic insulin aspart 30 at dinner in combination with metformin (500-2000 mg up to three times daily)
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 219 | 222
mmol/L
  Before Breakfast, N= 213, 213 | -2.52 (0.10) [-0.36 to 0.18] | -2.43 (0.10)
  2 hours After Breakfast, N= 213, 210 | -3.92 (0.17) [-0.38 to 0.55] | -4.00 (0.17)
  Before Lunch, N= 213, 210 | -2.80 (0.13) [-0.45 to 0.27] | -2.71 (0.13)
  2 hours After Lunch, N= 213, 211 | -4.37 (0.19) [-1.72 to -0.72] | -3.15 (0.18)
  Before Dinner, N= 212, 212 | -3.83 (0.16) [-1.41 to -0.58] | -2.83 (0.15)
  2 hours After Dinner, N= 211, 209 | -3.46 (0.18) [-0.58 to 0.41] | -3.37 (0.18)
  Bedtime, N= 207, 207 | -2.93 (0.15) [-0.24 to 0.55] | -3.09 (0.15)
  3:00 AM, N= 211, 210 | -1.99 (0.13) [-0.44 to 0.24] | -1.89 (0.13)
  Average, N= 213, 212 | -3.23 (0.10) [-0.55 to -0.03] | -2.94 (0.10)

4. Secondary Outcome: Change and Daily Average in Prandial Plasma Glucose Increment
Description: Change in prandial (mealtime) plasma glucose increment from baseline (week 0) to end of treatment (week 16). Daily average prandial plasma glucose increment was calculated at end of treatment.
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 219 | 222
mmol/L
  At Breakfast, N= 213, 210 | -1.41 (0.16) | -1.58 (0.16)
  At Lunch, N= 213, 210 | -1.57 (0.19) | -0.44 (0.19)
  At Dinner, N= 210, 209 | 0.40 (0.18) | -0.53 (0.18)
  Average, N= 213, 211 | -0.88 (0.11) | -0.84 (0.11)

5. Secondary Outcome: The Total Increase in Total Daily Insulin Dose Per Body Weight
Description: The total increase in total daily insulin dose per body weight from baseline (week 0) to end of treatment (week 16).
Time Frame: week 0, week 16
Population: Intention-to-Treat analysis set (ITT) is all randomised subjects exposed to at least one dose of trial product.
Measure: Least Squares Mean (Standard Error); unit: U/kg
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 210 | 210
U/kg | 0.963 (0.016) | 0.820 (0.015)

6. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to end of treatment (week 16)
Time Frame: week 0, week 16
Population: Intention-to-Treat analysis set (ITT) is all randomised subjects exposed to at least one dose of trial product.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 210 | 209
kg | 1.188 (0.157) | 0.817 (0.155)

7. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes occurring after baseline (week 0) to the end of treatment (week 16) in each treatment group. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no plasma glucose or blood glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-16
Population: Intention-to-Treat analysis set (ITT) is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 219 | 222
episodes
  All | 728 | 679
  Major or Minor | 158 | 198
  Minor | 157 | 198
  Symptoms Only | 570 | 481

8. Secondary Outcome: Number of Nocturnal Hypoglycaemic Episodes
Description: Number of nocturnal hypoglycaemic episodes occurring after baseline (week 0) to end of treatment (week 16) in each treatment group. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no plasma glucose or blood glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-16
Population: Intention-to-Treat analysis set (ITT) is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Number analyzed (Participants) | 219 | 222
episodes
  All | 134 | 81
  Major or Minor | 31 | 30
  Minor | 31 | 30
  Symptons Only | 103 | 51

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a time span of 16 weeks.
Description: Safety analysis set is all subjects exposed to at least one dose of trial product.
Arm/Group | BIAsp 50-50-30 | BIAsp 30-30
Serious Adverse Events (participants affected / at risk) | 5/219 | 9/222
Other Adverse Events (participants affected / at risk) | 74/219 | 68/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 50-50-30 (N=219) | BIAsp 30-30 (N=222)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 50-50-30 (N=219) | BIAsp 30-30 (N=222)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 10 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 (15) | 13 (13)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mucosal hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (2)
Injection site nodule (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (4)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vertebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Albumin urine present (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Manuscripts for publication will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications; however Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.